CLINICAL TRIAL: NCT05452369
Title: Ultrasound Guided Rhomboid Intercostal Nerve Block Versus Erector Spinae Plane Block for Postoperative Analgesia in Modified Radical Mastectomy:A Comparative Study
Brief Title: Postoperative Anelgesic Effect of Rhomboid Intercostal Nerve Block Versus Erector Spinae Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ghada fouad (Other)
Responsible Party: Sponsor-Investigator, ghada fouad, associate professor of anesthesia, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MFM-IRB,MS.21.09.1654
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Post Operative Pain
Keywords: Modified Radical Mastectomy; Rhomboid Intercostal Nerve Block; Erector Spinae Plane Block .
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: - Two arms: rhomboid intercostal plane block is the first group Erector spinae plane block is the second group
Who Masked: Participant, Outcomes Assessor
Masking Description: - double-blind comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rhomboid intercostal plane block (Experimental): as in intervention description
  Interventions: Drug: Rhomboid intercostal plane block
- Erector spinae plane block (Experimental): As in intervention description
  Interventions: Drug: Rhomboid intercostal plane block

INTERVENTIONS:
Drug: Rhomboid intercostal plane block — - 30 mL bupivacaine 0.25% will injected ultrasound-guided in rhomboid intercostal fascial plane .
  Other Names: fascial plane block

SUMMARY:
Despite of analgesic effect of intravenous analgesic medications at intraoperative and postoperative time , The regional anesthetic techniquehas more benefits suchbetter control of Acute pain and hence less chronic pain and decreases the need for opioids and analgesics to preserve immune function which responsible for higher rates of infection and local recurrence, even metastasis .

New regional anesthetic technique for modified radical mastectomy discovered recently called rhomboid intercostal nerve block that will compared against erector spinae plane block .

DETAILED DESCRIPTION:
The aim of this study is to compare the post-operative analgesic effect of ultrasound-guided rhomboid intercostal nerve block versus erector spinae plane block as regard total analgesic requirements, duration of effective analgesia,postoperative visual analog score (VAS), peri-operative hemodynamics,peri-operative complications and incidence of chronic postmastectomy pain.The technique of rhomboid intercostal nerve block:

After induction of anesthesia, the patient will be positioned in lateral decubitus with the operated side above. After sterilization of the patient's back, A linear ultrasound transducer (6-12 MHz) will place medial to the lower border of the scapula with the orientation marker directed cranially. The ultrasound landmarks, trapezius muscle, rhomboid muscle, intercostal muscles, pleura, and lung will be identified. The tissue plain between the rhomboid major and intercostal muscles is identified, and a single injection is administered at the T4-5. 80mm 21-gage needle will be inserted in the plane view of the ultrasound probe at the level of T4-5. After negative aspiration of blood or air, the rhomboid intercostal plane was hydro located with 2 mL of normal saline to confirm the correct needle tip position. A single injection of 30 ml of bupivacaine 0.25% will be applied into the interfacial plane between the rhomboid major and intercostal muscles. The spread of local anesthetic solution under the rhomboid muscle will be visualized by ultrasonography.

The technique of Erector spinae plane block (ESP):

After induction of anesthesia, the patient will be positioned in lateral decubitus with the operated side above. After sterilization of the patient's back, A linear ultrasound probe willplace 3-cm lateral to the midline at the level of T5 interspinous space and transverse process and three muscles willidentify: trapezius, rhomboid major, and erector spinae. A 10-cm needle was inserted craniocaudally in-plane, to reach the transverse process. After hydrodissection of the plane with 3 mL of normal saline, 30 ml of 0.25% bupivacainewilldeposit and thus erector spinae muscle will lift off the transverse process.

Block assessment will be performed using ice cube withtemperature of 4°C at midclavicular linein post anesthesia care unit after Full recovery which be confirmed when Aldrete's score ≥9 .

Block success means at least3 dermatomal segments should be having decreased sensation to cold.

Failed block will be excluded from the study and patient will replaced by another patient.

ELIGIBILITY:
Inclusion Criteria:

* - Female patients aged between 25-65 years.
* ASA physical status I or II.
* Scheduled for elective unilateral modified radical mastectomy

Exclusion Criteria:

* - Patient refusal.
* Infection at the site of injection.
* Hypersensitivity to the local anesthetic
* Bleeding disorders.
* Patients with cardiac, hepatic, and renal failure.
* BMI ≥40 kg/m2
* Patient with serum cr > 1.5

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients undergoing modified radical mastectomy surgery
Enrollment: 104 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The total analgesic requirements during the first 24 hours postoperative. | 0,2,4,6,8,10,12,16,20,24 hours postoperatively
  All patients will receive standard postoperative analgesia (1gm paracetamol every 8 hours IV).

SECONDARY OUTCOMES:
The duration of effective analgesia | 0,2,4,6,8,10,12,16,20,24 hours postoperatively
  time interval between the end of surgery and first analgesic request .

CONTACTS AND LOCATIONS:
Overall Officials: mohamed y makharita, MD, Study Director — Professor OFanesthesia Mansoura university; ghada f amer, MD, Study Chair — Assistant professor of anesthesia Mansoura university; ahmed E Kamal, resident, Principal Investigator — resident of anesthesia mansoura university
Locations (2):
- Egypt (2):
  - Mansoura University, Al Mansurah, Dakahlia Governorate
  - Mansoura University, Al Mansurah